CLINICAL TRIAL: NCT02652273
Title: Inhibition of Co-Stimulation in Rheumatoid Arthritis
Acronym: ICoSRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN13RH410; 2014-004419-35 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abatacept (Experimental): Abatacept 125mg administered via subcutaneous injection once a week for 24 weeks
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Abatacept 125mg/ml

SUMMARY:
The purpose of this study is to use abatacept as a clinical molecular probe to evaluate the effects of inhibiting costimulation on immune responses in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory immune mediated arthritis which leads to pain, swelling and destruction of joints. RA affects more than 500,000 subjects in the United Kingdom (UK) and incurs significant health and economic cost. Most patients require potent immune suppressing drugs such as methotrexate, which help reduce pain and stiffness, and protect the joints against damage. However, many patients do not respond or are unable to tolerate methotrexate. In these patients, biologic drugs such as abatacept are used to try to control the arthritis.

Abatacept is designed to target and inhibit a specific molecule involved in "costimulation" of the inflammatory signal that is thought to be important in RA. While abatacept has been shown to be effective in trials and clinical practice, the exact mechanism of action of abatacept in RA has not been fully elucidated. Understanding these actions is likely to inform both the use of abatacept in RA and lead to increased understanding of inflammation in humans with implications for further therapies. This six month prospective open label study, therefore, aims to investigate the effects of inhibiting costimulation on a variety of important inflammatory cell types and processes in humans with RA.

25 participants with RA who have bad prognostic genetic markers (Anti-citrullinated protein antibodies (ACPA) and human leukocyte antigen (HLADR4) and who were scheduled to receive subcutaneous abatacept as part of their standard clinical treatment will be recruited. Consenting participants will followed for a total of 24 weeks during which time they will have additional venous blood and urine samples taken to investigate the effects of abatacept on their immune cells and system. The primary endpoint of the study is the characterisation of the immune response following costimulatory modulation in RA patients at 12 weeks. Secondary endpoints include change in immunological response and its association with clinical outcome measures up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* RA as defined by the 2010 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria
* Eligible for abatacept therapy according to local/national guidelines

  * Active RA defined by DAS28 score required by local guidelines for eligibility for abatacept
  * Have previously failed (efficacy or tolerance) at least one disease-modifying antirheumatic drug (DMARD)
  * Have no contraindications to treatment with abatacept
* Be able to tolerate methotrexate at dose of 10-25mg/week, either orally or subcutaneously
* Anti-cyclic citrullinated peptide (CCP) positive
* Human leukocyte antigen D related (HLA-DR) B1*0401 or 0404) positive
* Able and willing to give written informed consent and comply with the requirements of the study protocol

Exclusion Criteria:

* History of or current autoimmune rheumatic disease other than RA
* Concomitant use of any biologic agent, including tumor necrosis factor (TNF) inhibitors
* Previous abatacept treatment
* Patients requiring >10mg prednisolone daily or intramuscular (IM) corticosteroids
* Active infection
* Known HIV or hepatitis B/C infection
* Latent tuberculosis (TB) infection
* Malignancy (other than non-melanoma skin cell cancers) within 5 years
* Women who are pregnant, women of childbearing potential who are unwilling to use appropriate contraception or breast-feeding
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Immunological response | Baseline and 12 weeks
  Change in T cell immune response to citrullinated peptides following costimulatory modulation

SECONDARY OUTCOMES:
Immunological response | Baseline, 4, 12 and 24 weeks
  Change in immunological response from baseline, as measured by transcriptional profile of relevant cell subset
Clinical response American College of Rheumatology (ACR) 20 | Baseline and 24 weeks
  Change in ACR 20 from baseline
Clinical response Disease Activity Score (DAS)28 | Baseline and 24 weeks
  Change in DAS 28 from baseline
T cell profile | Baseline, 12 and 24 weeks
  Change in T cell subpopulation profile from baseline
T cell response | 24 weeks
  Antigen-specific T cell response to tetanus
DC (CD11c+) phenotype | 24 weeks
  Dendritic cell (DC) (CD11c+) phenotype as measured by major histocompatibility complex (MHC) II expression
Biomarkers | 24 weeks
  Preliminary identification of biomarkers of response using urinary metabol/proteomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Iain McInnes, Prof, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne